CLINICAL TRIAL: NCT01021956
Title: A Phase IIa, Safety and Preliminary Effects Study of WST11 (Stakel®) Mediated Vascular-Targeted Photodynamic (VTP) Therapy in Subjects With Choroidal Neovascularization (CNV) Associated With Age-Related Macular Degeneration (AMD)
Brief Title: Safety and Preliminary Efficacy Study of WST11 (Stakel®)-Mediated VTP Therapy in Subjects With CNV Associated With AMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Retinal vascular occlusion in 2 patients
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN905 MLT202
Record Dates: First submitted 2009-11-29; First posted 2009-12-01 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: Macular Degeneration; Age Related Macular Degeneration; Choroidal Neovascularization; AMD; CNV; WST11; Stakel; Photodynamic therapy; Vascular Targeted Photodynamic therapy; VTP
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — padeliporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WST11 (STAKEL) (Experimental): Single doses of 2.5 mg/kg of STAKEL® in combination with transpupilar illumination of the macula at escalating doses from 12.5 to 75 Joules/cm².
  Interventions: Drug: STAKEL

INTERVENTIONS:
Drug: STAKEL — Open-label,safety and exploratory efficacy study in subjects with active CNV followed for 12 weeks.During first stage(dose escalating stage) subjects assigned to group 1 to 4 will receive a single treatment of VTP at one of three light levels and one of two Drug Light Interval (DLI).Second stage(dose confirmation)will be only initiated at a dose level in which an effect has been seen at week 1 and there is a maximum of one Dose Limiting Toxicity (DLT) out of three subject at week 5.
  Other Names: WST11

SUMMARY:
The objectives of this study are to evaluate the safety(first objective) and efficacy(second objective)of an experimental drug product,Stakel®, in the treatment of neovascular Age related Macular Degeneration (AMD). The drug product is activated in patients by exposure to light at a specific wavelength ("Vascular Targeted Photodynamic therapy", "VTP"). The exploratory objective is to assess whether it is possible to delay or reduce the requirement for anti Vascular Endothelium Growth Factor (anti VEGF) intravitreal therapy in the first 12 weeks after VTP.

All subjects will have a 52 weeks safety follow up telephone call (Not for Adverse Events (AEs) collection).

DETAILED DESCRIPTION:
The primary objective of this Phase IIa clinical study is to evaluate the safety of treatment with Stakel®-mediated VTP in subjects with neovascular AMD. The secondary objective of this Phase IIa clinical study is to explore the effect of treatment with Stakel®-mediated VTP in subjects with neovascular AMD. The exploratory objective is to assess whether it is possible to delay or reduce the requirement for anti Vascular Endothelium Growth Factor (anti VEGF) intravitreal therapy in the first 12 weeks after VTP.

All subjects will have a 52 weeks safety follow up telephone call. (Not for AEs collection).

ELIGIBILITY:
Inclusion Criteria:

* Twenty eight days or more after at least one ranibizumab injection, recurrent leakage on Fluorescein Angiography (FA) from subfoveal Choroidal NeoVessels (CNV) secondary to AMD.
* Total lesion size not exceeding 5400 μm in its greatest linear dimension.
* Best Corrected Visual Acuity (BCVA) letter score of 73 to 23 in the study eye at a starting distance of 4 meters.
* No contraindication to intravitreal ranibizumab injection.
* Postmenopausal for at least 12 months prior to enrollment or practicing medically acceptable form of birth control and not pregnant. Male subjects must be practicing a medically acceptable form of birth control.

Exclusion Criteria:

* Prior treatments:

  * Previous subfoveal laser photocoagulation, external-beam radiation therapy, or transpupillary thermoTherapy (TTT) in the study eye at any time.
  * Using anti-VEGF therapies for other indications (e.g., cancer) in the 30 days prior to the study and/or during the study
  * Received anti-VEGF injection in study eye during less than 28 days prior to Day 1 of the study.
  * More than three previous photodynamic therapy (PDT) treatments in the preceding 12 months.
  * Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within the preceding month.
  * History of vitrectomy,of glaucoma filtering surgery,submacular surgery or other surgical intervention in the study eye.
  * History of corneal transplant in the study eye.
  * Previous participation in any studies of investigational drugs within 1 month preceding Day 1 (excluding vitamins and minerals).
* Lesion Characteristics

  * Permanent structural damage to the center of the fovea of the study eye, or a concurrent ocular or systemic condition that could contraindicate administration of an investigational drug, or render the subject at a high risk of treatment complications.
  * Subretinal hemorrhage in the study eye that involves the center of the fovea, if the size of the hemorrhage is either ≥50% of the total lesion area or ≥1 disc area in size.
  * Subfoveal fibrosis or atrophy in the study eye which is at least 50% of the lesion.
  * CNV in either eye due to other causes.
  * Retinal pigment epithelial tear involving the macula in the study eye.
* Concurrent Ocular Conditions

  * Active intraocular inflammation (grade trace or above) or current vitreous hemorrhage or rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
  * History of idiopathic or autoimmune-associated uveitis in either eye.
  * Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
  * Aphakia or absence of the posterior capsule in the study eye.
  * Spherical equivalent of the refractive error in the study eye demonstrating more-than eight diopters of myopia.
  * Intraocular surgery (including cataract surgery) in the study eye within three months preceding Day 1.
  * Uncontrolled glaucoma in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bressler, Professor, Study Chair — Johns Hopkins University; Victor Gonzalez, Professor, Principal Investigator — Valley Retina Institute; John Wells, Professor, Principal Investigator — Palmetto Retina Center; Francine Behar Cohen, Professor, Principal Investigator — Hotel Dieu Hospital; Adrienne Scott, Doctor, Principal Investigator — Johns Hopkins/ Wilmer Eye Institute
Locations (4):
- United States (3):
  - Johns Hopkins,Wilmer Eye Institute, Baltimore, Maryland
  - Palmetto Retina Center, West Columbia, South Carolina
  - Valley Retina Institute, Harlingen, Texas
- Hotel Dieu de Paris Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No
The data are available in case report form for each patient

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1a -2.5 mg/kg STAKEL - 25 J/cm²: 2.5 mg/kg dose of STAKEL - 25 Joules/cm² of laser light at 753 nm
- Group 1b-2.5 mg/kg STAKEL - 12.6 J/cm²: 2.5 mg/kg dose of STAKEL -12.6 Joules/cm² of laser light at 753 nm
- Group 1c-2.5 mg/kg STAKEL - 18.9 J/cm²: 2.5 mg/kg dose of STAKEL -18.9 Joules/cm² of laser light at 753 nm
- Group 2-2.5 mg/kg STAKEL - 50 J/cm²: 2.5 mg/kg dose of STAKEL - 50 Joules/cm² of laser light at 753 nm
Period: Overall Study
Arm/Group | Group 1a -2.5 mg/kg STAKEL - 25 J/cm² | Group 1b-2.5 mg/kg STAKEL - 12.6 J/cm² | Group 1c-2.5 mg/kg STAKEL - 18.9 J/cm² | Group 2-2.5 mg/kg STAKEL - 50 J/cm²
Started | 3 | 3 | 3 | 1
Completed | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1a: 2.5 mg/kg - 25 Joules/cm²
- Group 1b: 2.5 mg/kg - 12.6 Joules/cm²
- Group 1c: 2.5 mg/kg - 18.9 Joules/cm²
- Group 2: 2.5 mg/kg - 50 Joules/cm²
- Total: Total of all reporting groups
Arm/Group | Group 1a | Group 1b | Group 1c | Group 2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.30 (7.51) | 78.3 (6.11) | 81.00 (6.08) | 87.00 (0) | 77.60 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 1 | 5
  Male | 3 | 0 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 3 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) - Number of Subjects With Eye Disorders
Description: Adverse events (AEs) consisting in Eye disorders, related or non related were collected throughout the study.
Time Frame: 12 week follow-up
Population: The safety analysis set included all subjects with a signed informed consent form who received study treatment
Measure: Number; unit: participants
Groups:
- Overall: All doses of TOOKAD Soluble and Laser Light
Arm/Group | Group 1a | Group 1b | Group 1c | Group 2 | Overall
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 10
participants | 3 | 1 | 0 | 1 | 5

2. Secondary Outcome: Visual Acuity
Description: Variation from baseline to week 12 in visual acuity score using Early Treatment Diabetic Retinopathy Study (ETDRS) 4.0 meter distance acuity chart.
  The patient is asked to read letter on a board from a distance of 4 meters. The charts use a geometric progression in letter size from line to line. The scores range from 0 (worse outcome) to 100/100 (best outcome)
Time Frame: Week 12.
Population: Although STAKEL® VTP procedure induced effective neovessels occlusion in some patients, as observed in the previous study (study MLT 2.01 ), due to the small number of patients treated and the early termination of the study, limited efficacy data is available and no efficacy conclusion can be drown from this study.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1a | Group 1b | Group 1c | Group 2
Number analyzed (Participants) | 3 | 3 | 3 | 1
score on a scale | 2 [-20 to 22] | -12 [-12 to 0] | 4 [-7 to 7] | -33 [-33 to -33]

3. Post Hoc Outcome: Number of Participants With Any Ocular or Non-ocular Adverse Events
Description: Global safety assessment including record of all complications and AEs, loss of lines in BCVA, slit lamp findings, IOP(Intra Occular Pressure), and fundus findings. All ocular and non-ocular AEs must be assessed for severity and relationship to the investigational product. Of note: the primary end point only concern patient with eye disorders events.
Time Frame: Day 1;Week 1;Week 5;Week 12.
Measure: Number; unit: participants
Arm/Group | Group 1a | Group 1b | Group 1c | Group 2
Number analyzed (Participants) | 3 | 3 | 3 | 1
participants | 3 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: systematic Assessment : Regular investigator assessment
Arm/Group | Group 1A | Group 1B | Group 1C | Group 2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 0/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1A (N=3) | Group 1B (N=3) | Group 1C (N=3) | Group 2 (N=1)
retinal vascular occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1A (N=3) | Group 1B (N=3) | Group 1C (N=3) | Group 2 (N=1)
eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Acuty reduced (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal pigment epitheliopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
macular ischaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less